CLINICAL TRIAL: NCT03312764
Title: Preventing Diabetes With Digital Health and Coaching for Translation and Scalability (PREDICTS)
Brief Title: Preventing Diabetes With Digital Health and Coaching
Acronym: PREDICTS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omada Health, Inc. (Industry)
Collaborators: University of Nebraska (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2017-03-06-001
Record Dates: First submitted 2017-10-06; First posted 2017-10-18 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: PreDiabetes
Keywords: Prediabetes; Obesity; Intensive behavioral counseling; Type 2 Diabetes
MeSH Terms: conditions — Prediabetic State; Obesity; Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to one of two groups for the duration of the study.
Who Masked: Investigator, Outcomes Assessor
Masking Description: All study investigators that collect data or analyze the data are prevented from knowing the interventions assigned to individual participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Diabetes Prevention Program (Experimental): Participants will receive access to a 12-month online diabetes prevention program modeled after the CDC DPP curriculum. Participants in the online program receive paced curriculum, access to a live health coach, interactive group message forums, and connected weight scale and activity monitoring devices.
  Interventions: Behavioral: Online diabetes prevention program
- Enhanced Standard Care (Active Comparator): All participants randomized to the standard-care/control group (SC) will be offered the opportunity to attend a single 90-minute diabetes prevention class with a trained health professional (MPH, RD, or related advanced degree). The class will focus on healthful eating based on the current MyPlate recommendations, guidance on gradual increases in moderate intensity physical activity, and action planning to be shared with friends and/or family. Control participants will also be given the opportunity to participate in the online digital intervention upon completion of the 12-month follow-up assessment.
  Interventions: Behavioral: Standard Care

INTERVENTIONS:
Behavioral: Online diabetes prevention program — Digital delivery of Intensive behavioral counseling for diabetes prevention and healthy lifestyle management. Recipients have access to online curriculum, a live health coach, group-based communication forums, and connected technology to track weight and physical activity.
  Arms: Online Diabetes Prevention Program
Behavioral: Standard Care — One-on-one or small group sessions with a dietitian or a trained health professional to advise on physical activity, healthful nutrition and risk reduction for diabetes.
  Arms: Enhanced Standard Care

SUMMARY:
The goal of this randomized controlled trial is to determine the efficacy of a digital diabetes prevention program for improving weight, glucose control, and secondary risk factors among people with prediabetes compared to an enhanced standard care plus wait-list control. Exploratory assessments of implementation facilitators and barriers will also be completed to determine strategies for integrating external diabetes-prevention interventions within healthcare settings.

DETAILED DESCRIPTION:
Prediabetes is an increasingly prevalent condition, characterized by glucose levels that are above normal but below the threshold for diabetes. Previous studies have demonstrated that intensive lifestyle interventions targeting changes in diet, physical activity, sleep, and stress can reduce the risk of progressing from prediabetes to Type 2 diabetes. The Diabetes Prevention Recognition Program (DPRP) currently recognizes both in-person and online programs that meet requirements to deliver approved curriculum, provide health coaching and group support, and equip participants with behavioral skills and self-monitoring tools to support behavior change. While non-randomized trial data demonstrate that an online digital program was successful for producing meaningful weight loss and improved glucose control, the goal of this randomized, controlled trial is to definitively evaluate the efficacy of the program for improving weight, glucose control and secondary risk factors compared to current standard care for prediabetes. In addition, few trials have examined the implementation factors that could speed the uptake of efficacious diabetes prevention interventions for delivery in regular clinical practice. Qualitative information on key organizational stakeholders (e.g., physicians, office managers) will be gathered to provide information on perceptions of the online program characteristics, outcomes, and resources concurrently with strategies to promote adoption and implementation in health care settings.

ELIGIBILITY:
Inclusion Criteria:

* Receives care at University of Nebraska Medical Center or Nebraska Medicine
* Age 19 years or older
* HbA1c 5.7%-6.4%
* Overweight (BMI 25+ or 22+ if Asian)
* Planning to reside in recruitment area for next 12 months
* Able to engage in moderate aerobic physical activity
* Medically stable
* Able to provide informed consent
* Willing to accept random assignment to treatment

Exclusion Criteria:

* Not meeting all inclusion criteria
* Diagnosed with Type I or II diabetes
* Diagnosed with congestive heart failure, coronary artery disease, chronic obstructive pulmonary disease, pulmonary hypertension
* Diagnosed with dementia or probable Alzheimer's disease
* Taking oral hypoglycemic agents
* Participating in a concurrent weight management program or interventional research protocol
* Unable to engage in physical activity
* On a prescribed medical diet
* Had bariatric surgery within the past 3 years or planning surgery within the next 12 months
* Anti-obesity or diabetes therapy within the preceding 4 months
* Any mental health condition, including eating disorders or alcohol/substance use, which would preclude full participation
* Self-report as currently pregnant or within 6 weeks of having given birth (or planning to become pregnant in the next 12 months)
* Unstable cardiac disease (i.e. heart attack/failure or stroke in the last 6 months, or in cardiac rehabilitation)
* On dialysis or an active organ transplant list
* Chronic kidney disease
* Untreated thyroid disease
* Cancer within the last 5 years unless skin cancer (i.e. currently or within the last 5 years in chemotherapy or radiation treatment)
* Unwilling to accept random assignment

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 598 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
HbA1c reduction | Baseline and 12 months
  Change in percent HbA1c

SECONDARY OUTCOMES:
Weight loss | Baseline, 4 months, and 12 months
  Reduction in percent of initial body weight
Decreased cardiovascular risk | Baseline, 4 months, and 12 months
  Atherosclerotic Cardiovascular Disease (ASCVD) risk estimator algorithm will be used to assess cardiovascular risk. The tool uses a number of demographic and health characteristics to estimate risk.

OTHER OUTCOMES:
Implementation Context | 12 months
  This qualitative assessment will identify the overall implementation climate for a digital DPP. Key informant interviews will be used to elicit stakeholder perceptions, which will be coded for meaning and grouped into categories. The categories will then be integrated to determine possible implementation strategies for this type of program. As such, there is a single assessment that will result in multiple categories. We identified the a priori hypothetical categories, but may find additional categories and may not find perceptions that align with the current categories. This is a single section since these qualitative outcomes may be variable.
  Physician, other health professional, and administrator perceptions of:
  1. The value and practicality of integrating a new DPP within their facility
  2. Barriers to DPP sustainability
  3. Contextual readiness for a diabetes prevention initiative
  4. Factors that would facilitate implementation
  5. Indicators of successful implementation

CONTACTS AND LOCATIONS:
Overall Officials: Paul Estabrooks, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual de-identified participant data that underlie the results reported in published manuscripts will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will be made available beginning 12 months and ending 36 months following article publication.
Access Criteria: Investigators who provide a methodologically sound proposal, and whose proposed use of the data has been approved by the Sponsor of the study will be given access to data. Data will be made available for participant data meta-analyses. Proposals should be directed to research@omadahealth.com. To gain access, requestors will need to sign a data access agreement. For approved proposals, data will be directly sent electronically to the requestor.

REFERENCES:
- [Derived] Katula JA, Dressler EV, Kittel CA, Harvin LN, Almeida FA, Wilson KE, Michaud TL, Porter GC, Brito FA, Goessl CL, Jasik CB, Sweet CMC, Schwab R, Estabrooks PA. Effects of a Digital Diabetes Prevention Program: An RCT. Am J Prev Med. 2022 Apr;62(4):567-577. doi: 10.1016/j.amepre.2021.10.023. Epub 2022 Feb 10. PMID 35151522